CLINICAL TRIAL: NCT02165319
Title: Comparison of the Cuff Pressure of an Endotracheal Tube After Supine-to-lateral Position Change: Barrel-shaped vs. Taper-shaped Cuff
Brief Title: The Cuff Pressure of an Endotracheal Tube After Supine-to-lateral Position Change
Acronym: LateralCuff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LateralTaperedCuff-phpkhc; LateralCuff_SNUH
Record Dates: First submitted 2014-05-27; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Intubation; Pain; Pharyngitis; Hoarseness; Cough
MeSH Terms: conditions — Pain; Pharyngitis; Hoarseness; Cough

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Barrel (Active Comparator): Endotracheal tube with barrel-shaped cuff will be used during general anesthesia.
  Interventions: Device: Barrel
- Tapered (Active Comparator): Endotracheal tube with tapered-shaped cuff will be used during general anesthesia.
  Interventions: Device: Tapered

INTERVENTIONS:
Device: Barrel — Barrel-shaped endotracheal tube will be used during general anesthesia.
  Arms: Barrel
Device: Tapered — Tapered-shaped tube will be used during general anesthesia.
  Arms: Tapered

SUMMARY:
To compare the cuff pressure in lateral position between barrel-shaped cuff and taper-shaped cuff

DETAILED DESCRIPTION:
The position of endotracheal tubes depends on the position of the patients. The change of the tube's position is known to influence the pressure of tube's cuff. The shape of the cuff (barrel-shaped versus tapered-shaped) may affect the tube's migration degree because of the difference of the frictional force.

The investigator try to compare the the cuff pressure after supine-to-lateral position change between barrel-shaped cuff and taper-shaped cuff.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for nephrectomy in lateral decubitus position

Exclusion Criteria:

* Pregnancy
* Patients with difficult airway
* Patients with neck motion disorder
* Patients with history of neck surgery
* Patients with history of oral and pharyngeal surgery
* Patients with body mass index > 35
* Patients without teeth

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
The cuff pressure after supine-to-lateral position change | At 10 minutes after anesthetic induction
  The cuff pressure will be measured after supine-to-lateral position change using the Manometer Portex®.

SECONDARY OUTCOMES:
The distance from the tube to the carina | At 10 minutes after anesthetic induction
  The distance from the tube to the carina will be measured using bronchoscopy after supine-to-lateral position change.
Complications related to endotracheal tube | At 0, 2, and 24 hours postoperatively
  Complications related to endotracheal tube (sore throat, hoarseness, dysphagia and cough) will be measured as 0:none, 1:mild, 2:moderate, 3:severe at 0, 2, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, PhD, Principal Investigator — Seoul National University of Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HC, Lee YH, Kim E, Oh EA, Jeon YT, Park HP. Comparison of the endotracheal tube cuff pressure between a tapered- versus a cylindrical-shaped cuff after changing from the supine to the lateral flank position. Can J Anaesth. 2015 Oct;62(10):1063-70. doi: 10.1007/s12630-015-0394-z. Epub 2015 Apr 17. PMID 25894912